CLINICAL TRIAL: NCT04644146
Title: Genetic Predisposition to Severe Forms of COVID-19 (SARS-CoV2 Infection) in Patients Without Comorbidities
Brief Title: Genetic Predisposition to Severe Forms of COVID-19 (SARS-CoV2 Infection)
Acronym: COVIDGEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1072
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: Coronavirus SARS CoV2; COVID-19; genetics; predisposition; critical care
MeSH Terms: conditions — COVID-19; Disease Susceptibility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA samples has been extracted for whole exome sequencing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SEVERE: Patients affected by SARS-CoV2 infection with severe lung dysfunction needing oxygen complementation and critical care supports - criteria 18-70yr old and without any comorbidities
  Interventions: Genetic: GENETIC
- CONTROL: Patients affected by SARS-CoV2, as shown by PCR and/or antigen testing diagnosis and without any or minor clinical expression
  Interventions: Genetic: GENETIC

INTERVENTIONS:
Genetic: GENETIC — It is a retrospective study on patients which has been hospitalized since the beginning of the COVID-19 pandemic in Lyon (march 2020). The blood samples have been collected I the frame of the regular follow-up of the patients and DNA extracted and conserved for the various research protocols ongoing in the University Hospital. The DNA will be analyzed by next generation sequencing

SUMMARY:
The main objective of this part of the project is to identify the germline genetic factors which discriminate the benign and severe forms of SARS-CoV2 (CoVID-19) infection in the context of the ongoing SARS-CoV2 (HCOVID-19) epidemic. The scientific arguments of the project are described in APPENDIX. We hypothesize that pathogenic variants in genes coding for crucial factors involved in the HOST PATHOGEN interaction could explain the susceptibility of some patients to severe disease, even in the absence of comorbidities. The challenge is to identify those of the genetic factors who may be related respiratory distress and potentially further death. Based on our previous experience in sarcoidosis, a multifactorial disease predisposing to opportunistic infections, we will focus particularly the regulation of apoptosis and autophagy, immune response to viral infection, and endoplasmic reticulum stress response (ER STRESS) which is closely linked to apoptosis. Genetic defects in such pathways may decrease the clearance of viral particles and induces the progressive invasion by SARS-CoV2 and destruction of lung parenchyma. Our strategy will be similar to that described in our previous studies on sarcoidosis, recently published. We will combine a comparative genotype analysis by WHOLE EXOME SEQUENCING (WES) of benign and severe forms of SARS-CoV2 infection through clinical subgroups defined by the infectious diseases experts and a bioinformatics analysis of the functional networks identified by the panel of genes sharing pathogenic variants and discriminating the severe forms of the diseases. WES data will be carefully analyzed and related to all the intracellular physiological process and also the functional pathways involved in host-pathogen interaction: viral targets on the cell surface and downstream signaling, viral genomic RNA replication and translation, production and release of new viral particles. Finally, our main objectives are the definition of a gene panel more specifically related to severe forms of infection and the characterization of defective pathways involved in pejorative forms of SARS-COv2 disease in order to identify putative therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by COVID-10 Age: 18-70 (values included) Without any co morbidities (analysis of the clinical files in our hospital) Without any regular treatments

Exclusion Criteria:

* below 18yr and higher than 70yr old
* With comorbidities - ex: diabetes, obesity, hypertension, ischemic heart, neurological disorders, autoinflammatory / autoimmune diseases …
* Not agreeing the protocol (absence of informed consent)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by COVID-10 Age: 18-70 (values included) Without any co morbidities (analysis of the clinical files in our hospital) Without any regular treatments
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary criteria of data evaluation | through study completion, average 6 months
  Number of genes affected by pathogenic variants in the SEVERE GROUP and for which no mutations have been observed in the CONTROL group For each gene sharing variants in the SEVERE GROUP and not in CONTROLS, the protein encoded by this gene will be identified and his function analyzed in the frame of various protein network software. The frequency of each mutation, so called the minor allele frequency will be evaluated in order to highlight only those which are rare (MAF < 0,01) in the normal population and thus suggesting a putative pathogenic role in the response to SARS-CoV2 infection.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital LYON (Hospices Civils de LYON), Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided